CLINICAL TRIAL: NCT05882539
Title: Construction of Risk Prediction Model for Oral Mucosal Pressure Injury in ICU Patients With Oral Tracheal Intubation
Brief Title: Oral Mucosal Pressure Injury in ICU Patients With Oral Tracheal Intubation
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Second Affiliated Hospital, School of Medicine, Zhejiang University (Other)
Responsible Party: Sponsor
Other Study IDs: 2022-0586
Record Dates: First submitted 2023-05-21; First posted 2023-05-31 (Actual); Last update posted 2023-05-31 (Actual); Status verified 2023-05

CONDITIONS: Oral Mucosal Pressure Injury
Keywords: Intensive Care Units; Intubation, Intratracheal; Mucosal Pressure Injury; Prediction Model
MeSH Terms: interventions — Constraint Induced Movement Therapy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 2 Weeks
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (10):
- endotracheal tube material: One group of patients used a spring-loaded endotracheal tube and the other group used a PVC tube.
  Interventions: Device: endotracheal tube material,Bite block Material
- Bite block Material: One group of patients used hard bite block and the other group used soft bite block
  Interventions: Device: endotracheal tube material,Bite block Material
- Moisture of oral mucosa: One group of patients had moist oral mucosa after entering the ward and the other group had dry oral mucosa.
  Interventions: Device: endotracheal tube material,Bite block Material
- serum albumin level: One group of patients had normal serum albumin level at the first blood sample analysis after tracheal intubation and the other group was abnormal.
  Interventions: Device: endotracheal tube material,Bite block Material
- mean arterial pressure level: One group of patients had normal mean arterial pressure leve after entering the ward and the other group was abnormal.
  Interventions: Device: endotracheal tube material,Bite block Material
- blood lactate level: One group of patients had normal blood lactate levels at the first blood sample analysis after tracheal intubation and the other group was abnormal.
  Interventions: Device: endotracheal tube material,Bite block Material
- constraint: One group of patients was constrained during follow-up and the other group was not constrained.
  Interventions: Device: endotracheal tube material,Bite block Material
- sedation: One group of patients was sedated during follow-up and the other group was not sedated.
  Interventions: Device: endotracheal tube material,Bite block Material
- prone position: One group of patients had a prone position performed during follow-up and the other group did not.
  Interventions: Device: endotracheal tube material,Bite block Material
- Duration of tracheal intubation: Dichotomous grouping of the duration of tracheal intubation according to the results of the study.
  Interventions: Device: endotracheal tube material,Bite block Material

INTERVENTIONS:
Device: endotracheal tube material,Bite block Material — Exposure factors associated with tracheal intubation in patients that may influence the occurrence of oral mucosa pressure injurie, such as the material and fixation of the tracheal tube, the patient's own nutrition, the level of tissue perfusion and relevant treatment factors.
  Other Names: Moisture of oral mucosa; serum albumin level; mean arterial pressure level; blood lactate level; constraint; sedation; prone position; Duration of tracheal intubation

SUMMARY:
In this study, based on the conceptual framework of Pressure Injurie development, the risk factors for pressure injury in critically ill patients provided by the latest guidelines, and combined with the current relevant studies on mucosal pressure injury, we prospectively observed and collected clinical data related to tracheal intubation patients in the ICU, analyzed the risk factors for the occurrence of oral MPI, and established a risk prediction model to help clinical and nursing staff to detect and actively prevent oral MPI at an early stage The study aims to improve the quality of nursing management, enhance the level of nursing services and improve patient satisfaction.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 18 years;
2. Duration of ICU admission ≥ 48h.

Exclusion Criteria:

1. radiotherapy oral mucositis;
2. Pressure injury to the mucosa, oral ulcers and erosions from other causes already present prior to tracheal intubation;
3. Patients undergoing oral surgery;
4. those who have been brought in from outside the hospital for >48h for transoral tracheal intubation;
5. Common oral ulcers (not pressure/friction generated).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: ICU patient with tracheal intubation inserted through the mouth
Sampling Method: Non-Probability Sample
Enrollment: 471 (Estimated)
Dates: Start 2023-01-01 (Actual); Primary Completion 2023-12-30 (Estimated); Study Completion 2024-12-30 (Estimated)

PRIMARY OUTCOMES:
oral mucosal pressure injury | up to 2 weeks
  Whether oral mucosal pressure injury occurred during the follow-up period

CONTACTS AND LOCATIONS:
Overall Officials: Zhu Yi Rong, Study Director — 2nd Affiliated Hospital, School of Medicine, Zhejiang University, China; Sun Yan, Principal Investigator — 2nd Affiliated Hospital, School of Medicine, Zhejiang University, China; Xiang Yan, Principal Investigator — 2nd Affiliated Hospital, School of Medicine, Zhejiang University, China; Guo Jingjing, Principal Investigator — 2nd Affiliated Hospital, School of Medicine, Zhejiang University, China
Locations (1):
- 2nd Affiliated Hospital, School of Medicine, Zhejiang University, Hangzhou, Zhejiang, China